CLINICAL TRIAL: NCT05482360
Title: Testing Implementation Strategies to Improve Delivery of Pre-exposure Prophylaxis (PrEP) for Pregnant and Postpartum Women in Kenya (K01)
Brief Title: Testing Implementation Strategies to Improve Delivery of PrEP for Pregnant and Postpartum Women in Kenya
Acronym: PrEPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anjuli Wagner, Assistant Professor, Global Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00008392-A; K01MH121124 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pre-Exposure Prophylaxis; HIV Infections; Pregnancy Related
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A difference-in-difference design will be used; this is a quasi-experimental design that compares data before an intervention is introduced to data after the intervention is introduced and compares that with the expected change before and after in comparison clinics. Three rounds of difference-in-differences tests will be used to evaluate three PrEP optimization interventions, identified by stakeholders based on qualitative information. Each of the three rounds will include 4 facilities receiving the intervention and 4 facilities serving as an ongoing concurrent comparator group; these 4 facilities will not receive any of the packages of interventions, but will undergo the same data collection procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Package 1 (Experimental): Package 1: Three implementation strategies including fast tracking, provider re-training, and dispensing PrEP in MCH
  Interventions: Other: PrEP Optimization Interventions
- Comparator for Package 1 (No Intervention): 4 facilities were assigned to the comparator group and never received any implementation strategy.
- Package 2 (Experimental): Package 2: Three implementation strategies including task shifting PrEP counseling from clinicians/nurses to HIV testing services providers (HTS), training different cadres, and dispensing PrEP in MCH
  Interventions: Other: PrEP Optimization Interventions
- Package 3 (Experimental): Package 3: Three implementation strategies including use of PrEP educational materials, PrEP health talks in waiting bays and dispensing PrEP in MCH
  Interventions: Other: PrEP Optimization Interventions
- Comparison for Package 2 (No Intervention): 4 facilities were assigned to the comparator group and never received any implementation strategy.
- Comparison for Package 3 (No Intervention): 4 facilities were assigned to the comparator group and never received any implementation strategy.

INTERVENTIONS:
Other: PrEP Optimization Interventions — There were three bundles of strategies tested determined based on the qualitative information gathered in Aim 1 by stakeholders
  Arms: Package 1; Package 2; Package 3

SUMMARY:
This study tests strategies for improving PrEP implementation in maternal and child health clinics using an interrupted time series.

DETAILED DESCRIPTION:
This study aims to improve integrated delivery of PrEP to women seeking health services in maternal and child health clinics by piloting and evaluating four strategies or bundles of strategies for optimized PrEP delivery. Strategies to be tested include three packages of strategies identified by stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving Maternal and Child Health (MCH) services HCW participating in satisfaction surveys

Exclusion Criteria:

* Unwilling or unable to provide informed consent

Ages: 15 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Anyone presenting for maternal child health services can be included in the study.
Enrollment: 5173 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjuli Wagner, PhD, Principal Investigator — University of Washington
Locations (1):
- Ober Health Center, Homa Bay, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the protocol section (5,173) includes the sum of participants who started in the participant flow module below (4,972), as well as the 201 additional health care workers who provided cross-sectional data in the intervention group during the intervention period. There was no drop-off between consent and enrollment.
Units Other Than Participants: Facilities
Groups:
- Comparator for Package 1; Comparator for Package 2; Comparator for Package 3: 4 facilities were assigned to the comparator group and did not receive any implementation strategies.
Period: Baseline Period (3 Months)
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Started | 392; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 420; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 402; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 415; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 419; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 406; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.)
Completed | 392; 4 Facilities | 420; 4 Facilities | 402; 4 Facilities | 415; 4 Facilities | 419; 4 Facilities | 406; 4 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities
Period: Intervention Period (3 Months)
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Started | 408; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 416; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 439; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 426; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 420; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 409; 4 Facilities
Completed | 408; 4 Facilities | 416; 4 Facilities | 439; 4 Facilities | 426; 4 Facilities | 420; 4 Facilities | 409; 4 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3 | Total
Number analyzed (Participants) | 392 | 420 | 402 | 415 | 419 | 406 | 2454
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 28] | 25 [22 to 29] | 23.5 [21 to 28] | 24 [22 to 29] | 24 [21 to 27] | 24 [21 to 29] | 24 [21 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 392 | 420 | 402 | 415 | 419 | 406 | 2454
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 392 | 420 | 402 | 415 | 419 | 406 | 2454
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 392 | 420 | 402 | 415 | 419 | 406 | 2454

OUTCOME MEASURES:

1. Primary Outcome: Change in PrEP Penetration
Description: Proportion of women who are screened for PrEP / total women receiving antenatal or postnatal services
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 800 | 836 | 841 | 841 | 839 | 815
Participants
  Baseline: number analyzed (Participants) | 392 | 420 | 402 | 415 | 419 | 406
  Baseline | 13 | 23 | 35 | 3 | 49 | 23
  Intervention: number analyzed (Participants) | 408 | 416 | 439 | 426 | 420 | 409
  Intervention | 23 | 7 | 93 | 22 | 146 | 27

2. Primary Outcome: Change in PrEP Fidelity
Description: Proportion of women who receive all PrEP specific steps in a visit: HIV testing, HIV risk screening, PrEP counseling. Assessed among the subset of women who are due for an HIV test, as per Kenyan guidelines, which is a subset of the overall sample.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 327 | 322 | 365 | 342 | 309 | 299
Participants
  Baseline: number analyzed (Participants) | 179 | 163 | 174 | 172 | 161 | 136
  Baseline | 9 | 8 | 15 | 1 | 23 | 14
  Intervention: number analyzed (Participants) | 148 | 159 | 191 | 170 | 148 | 163
  Intervention | 9 | 2 | 55 | 8 | 61 | 8

3. Primary Outcome: Timeliness of Services
Description: Time (minutes) spent receiving services from health care workers
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 384 | 384 | 383 | 384 | 384 | 384
minutes
  Baseline: number analyzed (Participants) | 192 | 192 | 191 | 192 | 192 | 192
  Baseline | 15 [10 to 29] | 14 [9.5 to 26.5] | 13 [9 to 23] | 12 [8 to 21] | 14 [8 to 29] | 15 [10 to 29]
  Intervention: number analyzed (Participants) | 192 | 192 | 192 | 192 | 192 | 192
  Intervention | 15 [10 to 31.5] | 12 [8.5 to 21.5] | 13 [9 to 22] | 15 [10.5 to 26] | 15 [10.5 to 28.5] | 15 [10 to 29]

4. Primary Outcome: Waiting Time
Description: Time (minutes) spent waiting to receive services
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 384 | 384 | 383 | 384 | 384 | 384
minutes
  Baseline: number analyzed (Participants) | 192 | 192 | 191 | 192 | 192 | 192
  Baseline | 47 [22 to 77.5] | 33 [13. to 57.5] | 37 [18 to 66] | 33 [14.5 to 63] | 47 [22 to 81] | 32.5 [16 to 69]
  Intervention: number analyzed (Participants) | 192 | 192 | 192 | 192 | 192 | 192
  Intervention | 42.5 [28 to 64] | 38 [14.5 to 73] | 43 [25 to 66.5] | 31.5 [15 to 56] | 35.5 [23 to 58] | 35 [14 to 71.5]

5. Primary Outcome: HCW Acceptability
Description: Total on 4 item Acceptability of Intervention Measures (AIM) score, 1 (Completely disagree) to 5 (Completely Agree) Likert scale. The minimum score on the 4 items is 4 points (scoring 1 on each of the 4 items) while the maximum is 20 points (scoring 5 on each of the 4 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: This outcome was assessed on a group of HCW who were involved in delivering the implementation strategy package. These are not a subset of the women enrolled in the study, hence the numbers are not concordant.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Package 1 | Package 2 | Package 3
Number analyzed (Participants) | 64 | 92 | 45
units on a scale | 18.5 [16 to 20] | 18 [16 to 20] | 20 [18 to 20]

6. Primary Outcome: Health Care Worker (HCW) Appropriateness
Description: Total on 4 item Intervention Appropriateness Measure (IAM) score, 1 (Completely disagree) to 5 (Completely Agree) Likert scale. The minimum score on the 4 items is 4 points (scoring 1 on each of the 4 items) while the maximum is 20 points (scoring 5 on each of the 4 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Package 1 | Package 2 | Package 3
Number analyzed (Participants) | 64 | 92 | 45
units on a scale | 18 [16 to 20] | 19 [16 to 20] | 20 [17 to 20]

7. Primary Outcome: Client Satisfaction
Description: Total on 7 item exit survey of clients to assess their satisfaction with services received at the facility, 1 (worse) to 4 (better) scale. The minimum score on the 7 items is 7 points (scoring 1 on each of the 7 items) while the maximum is 24 points (scoring 4 on each of the 7 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 800 | 836 | 841 | 841 | 839 | 815
units on a scale
  Baseline: number analyzed (Participants) | 392 | 420 | 402 | 415 | 419 | 406
  Baseline | 22 [20 to 23] | 22 [20 to 23] | 21 [20 to 22] | 20 [20 to 22] | 22 [20 to 23] | 21 [20 to 23]
  Intervention: number analyzed (Participants) | 408 | 416 | 439 | 426 | 420 | 409
  Intervention | 21 [20 to 22] | 21 [20 to 22] | 21 [20 to 22] | 21 [20 to 22] | 22 [21 to 23] | 22 [20 to 23]

8. Secondary Outcome: PrEP Uptake
Description: Proportion of women who accept PrEP among those offered
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
  This analysis population is a subset of the total because it only includes those who were offered PrEP, as noted in the denominator description of the indicator.
Measure: Count of Participants; unit: Participants
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 32 | 31 | 77 | 23 | 107 | 35
Participants
  Baseline: number analyzed (Participants) | 12 | 24 | 14 | 5 | 32 | 18
  Baseline | 2 | 2 | 2 | 0 | 7 | 4
  Intervention: number analyzed (Participants) | 20 | 7 | 63 | 18 | 75 | 17
  Intervention | 2 | 3 | 15 | 5 | 11 | 4

9. Secondary Outcome: PrEP Continuation
Description: Proportion of women who present for a refill among those initially prescribed PrEP
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
  This analysis population is a subset of the total because it only includes those who were initially prescribed PrEP, as noted in the denominator description of the indicator.
Measure: Count of Participants; unit: Participants
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 32 | 31 | 77 | 23 | 107 | 35
Participants
  Baseline: number analyzed (Participants) | 12 | 24 | 14 | 5 | 32 | 18
  Baseline | 2 | 6 | 2 | 0 | 5 | 8
  Intervention: number analyzed (Participants) | 20 | 7 | 63 | 18 | 75 | 17
  Intervention | 6 | 1 | 15 | 5 | 9 | 5

10. Secondary Outcome: Client PrEP Knowledge
Description: Number of participants with perfect knowledge on PrEP information questions based on content covered in counseling sessions
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 800 | 836 | 841 | 841 | 839 | 815
Participants
  Baseline: number analyzed (Participants) | 392 | 420 | 402 | 415 | 419 | 406
  Baseline | 3 | 6 | 0 | 0 | 0 | 0
  Intervention: number analyzed (Participants) | 408 | 416 | 439 | 426 | 420 | 409
  Intervention | 3 | 1 | 1 | 2 | 0 | 0

11. Secondary Outcome: PrEP Adherence
Description: Proportion of women who have >80 percent adherence to PrEP by pill count among those initially prescribed PrEP
Time Frame: 6 months
Population: During preparatory activities for data collection, it was determined that it was not feasible to extract patient adherence information,; this outcome was neither collected nor compared. It was not feasible to extract patient adherence information because routine program data at each facility different substantially in how it quantified adherence to PrEP; it was not possible, nor meaningful to collect or analyze these data.
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Package 3 | Comparison for Package 2 | Comparison for Package 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: PrEP Efficiency
Description: Patient flow mapping to identify more efficient client flows with fewer transitions between physical spaces and providers
Time Frame: 6 months
Population: During preparatory activities for data collection, it was determined that it was not feasible to collect efficiency. This outcome was neither collected nor compared. It was not feasible to quantify efficiency in the way in which we originally envisioned due to the heterogeneity between sites and within sites on how service provision was organized and delivered.
Units Other Than Participants: Facility
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
Number analyzed (Facility) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 cross-sectional visit. In this cross-sectional study, there were no participants followed longitudinally. Adverse events were not collected systematically within this minimal risk, cross-sectional study.
Arm/Group | Package 1 | Comparator for Package 1 | Package 2 | Comparator for Package 2 | Package 3 | Comparator for Package 3
All-Cause Mortality (participants affected / at risk) | 0/800 | 0/836 | 0/841 | 0/841 | 0/839 | 0/815
Serious Adverse Events (participants affected / at risk) | 0/800 | 0/836 | 0/841 | 0/841 | 0/839 | 0/815
Other Adverse Events (participants affected / at risk) | 0/800 | 0/836 | 0/841 | 0/841 | 0/839 | 0/815

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT05482360/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT05482360/ICF_001.pdf